CLINICAL TRIAL: NCT03658096
Title: Quantitative Assessment of Distal Radioulnar Joint Stability With Pressure-Monitor Ultrasonography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tokyo Medical University (Other)
Responsible Party: Principal Investigator, Yuichi Yoshii, Associate Professor, Department of Orthopaedic Surgery, Tokyo Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 17-26
Record Dates: First submitted 2018-08-27; First posted 2018-09-05 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Distal Radioulnar Joint Sprain; Triangular Fibrocartilage Complex Injury

STUDY DESIGN:
Intervention Model Description: patients and healthy controls
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy volunteer (Active Comparator)
  Interventions: Device: pressure monitor ultrasound system
- DRUJ instability patients (Active Comparator)
  Interventions: Device: pressure monitor ultrasound system

INTERVENTIONS:
Device: pressure monitor ultrasound system — Patients and healthy volunteers will be tested sitting with the elbow flexed and the forearm pronated. The forearm of the examinee will be secured to the table. The hand will be positioned on an adjustable block such that the forearm will be in a horizontal position. At the distal radioulnar joint level, the transducer will be maintained perpendicular to the longitudinal axis of the ulna. The dorsal surface of the distal radius and the center of the ulnar head will be displayed on a monitor.To determine the same measurement level in each volunteer, the highest aspect of the ulnar head will be taken. The DRUJ motion during cyclic loading toward the palmar direction at the distal ulna will be recorded. The compression-release cycles will be applied with the pressure-monitor ultrasound system. The cycle will be set to 1.5Hz. The pressure in the palmar direction will be applied with different levels of transducer displacements, i.e. 1 mm, 2 mm, and 3 mm.

SUMMARY:
To quantitatively assess distal radio ulnar joint (DRUJ) stability, a pressure-monitor ultrasound system was developed. The objective of this study was to evaluate the force-displacement relationship of DRUJ in patients and normal subjects. Each subject will be imaged sitting with elbow flexed and forearm pronated. The dorsal surface of distal radius and the center of ulnar head will be displayed at DRUJ level. The pressure toward palmar direction will be applied to distal ulna with different levels of transducer displacements, i.e. 1 mm, 2 mm, and 3 mm. The distance between the dorsal surface of the ulnar head and the dorsal surface of the distal radius will be measured. At the same time, the pressure to the transducer will be measured.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* DRUJ instability patients

Exclusion Criteria:

* the participants who had a history of previous wrist trauma and wrist pain will be excluded

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2024-08-27 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Instability of distal radioulnar joint (pressure) | 1 year
  According to the measurements of the pressure to distal radioulnar joint, determine if the exam can distinguish patients from healthy subjects.
Instability of distal radioulnar joint (dsiplacement) | 1 year
  According to the measurements of the displacement of distal radioulnar joint, determine if the exam can distinguish patients from healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Tomoo Ishii, Study Director — Tokyo Medical University Ibaraki Medical Center
Locations (1):
- Tokyo Medical University Ibaraki Medical Center, Ami, Ibaraki, Japan

IPD SHARING:
Plan to Share IPD: No